CLINICAL TRIAL: NCT03531125
Title: A Phase 0, Pre-operative, Window-of-opportunity Study to Assess Gene Expression in Patients With Resectable, Locally Advanced, or Metastatic Pancreatic Cancer (NEOPANC-01)
Brief Title: Gene Expression in Pancreatic Cancer
Acronym: NEOPANC-01
Status: Terminated | Type: Observational
Why Stopped: Study was closed early due to low numbers of evaluable patients
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OCTO_087
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Tumour biopsy
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic Ultrasound — Endoscopic ultrasound for tumour biopsy collection
Procedure: Pancreaticoduodenectomy — Surgery to remove pancreatic tumour

SUMMARY:
Pancreatic cancer is a lethal disease. The 1-year and 5-year survival rate is approximately 20% and <5% respectively. The treatment options available are limited. Only around 10-20% of patients present early enough to undergo surgical resection. Furthermore, chemotherapy for more advanced pancreatic cancer leads to limited survival benefit and can cause significant side effects. One of the main obstacles to developing new treatments for pancreatic cancer is the limited understanding of how pancreatic cancer cells change/evolve/adapt following treatment.

This study is a pilot study to assess whether the investigators can track gene expression (using a technique called RNA sequencing) in pancreatic cancer cells between two separate time points. Investigators intend to take a tissue sample (biopsy) of the cancer using endoscopy ultrasound (EUS) and compare it with samples taken either at the time of surgery in those patients with resectable disease or follow-up EUS derived biopsies in irresectable cancers.

The interval between endoscopy and follow-up EUS or surgery will be approximately 2 to 3 weeks and reflects the standard period of time that patients wait from the time point at which the cancer is deemed to be operable (in the multi-disciplinary team meeting) to the actual operation.

If the investigators find that the samples (biopsies) taken at EUS and at surgery or follow-up EUS are comparable they plan to develop future clinical trials of similar design but with the addition of drug therapy. The investigators will use RNA sequencing to interrogate the effects of novel cancer drugs on gene expression within the tumour. This will give them information on how to select patients for therapy, how resistance develops to these treatments, and allow the investigators to better understand what treatments can be combined on a rational basis. However, prior to undertaking such studies it is important to understand how much variability there is in gene expression between sampling at 2 different time points at which two different techniques are used.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, aged 18 years or above
2. Patients with pancreatic cancer planned for surgical resection, or patients with locally advanced or metastatic pancreatic cancer
3. For patients planned for resection the tumour must be within the head of the pancreas such that the EUS biopsy sites and needle track can be resected surgically
4. Adequate blood clotting parameters in order to undergo an EUS with biopsies, evidenced by the following:

   1. Platelet count ≥ 75 x 109L
   2. International normalised ratio (INR) ≤ 1.5
5. Patients have given written informed consent and are willing and able to comply with the scheduled visits, laboratory tests and study procedures including endoscopy (e.g. patients able to lie flat without being breathless and have no evidence of oesophageal stricture)

Exclusion criteria:

1. Previous histologically or cytologically confirmed pancreatic tumour that is not adenocarcinoma
2. Other psychological, social or medical condition, physical examination finding(s) or a laboratory abnormality that the investigator(s) considers would make the patient a poor study candidate or could interfere with protocol compliance or the interpretation of study results
3. Positive screening pregnancy test if woman of child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of whole transcriptome RNA sequencing of EUS derived pre-operative sample and whole transcriptome RNA sequencing of biopsies either taken from the pancreatic cancer during resection or repeat biopsy using EUS | Up to 6 weeks - Time between Endoscopic Ultrasound and surgery or follow up EUS

SECONDARY OUTCOMES:
Percentage and number of patients that undergo EUS and follow up EUS or surgery that have a) histopathological evidence of adenocarcinoma in their biopsy and surgical samples, and b) of suitable RNA quality for analysis | Up to 6 weeks - Time between Endoscopic Ultrasound and surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom